CLINICAL TRIAL: NCT02489955
Title: Prospective Randomised Trial of 'Area Under the Curve' (AUC) Dosing Strategy for Intravenous Tobramycin Versus Standard Trough Dosing for Pulmonary Exacerbations in Adult Patients With Cystic Fibrosis (CF)
Brief Title: Antibiotic Nephrotoxicity in Adult Patients With Cystic Fibrosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Leeds Teaching Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RM14/11283
Record Dates: First submitted 2015-05-18; First posted 2015-07-03 (Estimated); Last update posted 2015-07-03 (Estimated); Status verified 2015-07

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — Amikacin; Tobramycin

ARMS (2):
- AUC group (Experimental)
  Interventions: Drug: Amikacin; Drug: Colomycin
- Trough dose monitoring (Active Comparator)
  Interventions: Drug: Tobramycin

INTERVENTIONS:
Drug: Amikacin
  Arms: AUC group
Drug: Tobramycin
  Arms: Trough dose monitoring
Drug: Colomycin
  Arms: AUC group

SUMMARY:
Adult patients with cystic fibrosis (CF) are treated with high dose antibiotics to reduce the long term damage to their lungs from infection. This would typically be with a two week course of intravenous antibiotics each time they have a chest infection (typically three to four times a year).

The most effective and commonly used antibiotic in most cases is tobramycin. If this cannot be used because of previous side effects, allergy or a resistant infection then colomycin or amikacin are usually used. Each of these antibiotics are known to be toxic to both the kidneys and ear. As patients are living longer (into their forties), the total amount of these antibiotics they are receiving over their lifetime is increasing. This is now leading to increased complications such as kidney damage and hearing loss. Because of this, the investigators need to look at methods to accurately quantify damage and reduce potential kidney and hearing damage.

The investigators intend to quantify kidney damage by measuring new protein markers within the urine and blood that signify kidney damage before more conventional and currently available methods are able to.In those patients treated with intravenous tobramycin the investigators will also look at an alternative method used to calculate the most appropriate dose of antibiotic for each participant. This dosing method is called 'area under the curve or AUC' dose monitoring. This method currently in clinical use in other countries is thought to more accurately reflect the most appropriate dose for each participant and thus reduce the chance of kidney and hearing problems. This 'AUC' method requires two rather than one dose level to be checked each time a dose calculation is made. Participants receiving tobramycin will be randomised to receive dosing by this method or the investigators' currently used method of 'trough' monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CF*
* Able to give written informed consent
* Pulmonary exacerbation requiring IV tobramycin, amikacin or colistin based on the decision of the treating physician

Exclusion Criteria:

* Known allergy or adverse reaction to proposed antibiotic (tobramycin, amikacin or colistin)
* Pregnancy (if found to be pregnant during the study the participant will be immediately withdrawn)
* Continuation of nebulised aminoglycoside or colistin during IV treatment
* Use or intended use of NSAIDS

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2015-02; Primary Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
Area Under the Curve' (AUC) of tobramycin | Days 1, 8, 14, 28
Area Under the Curve' (AUC) of Amikacin or Colomycin | Days 1, 8, 14, 28

CONTACTS AND LOCATIONS:
Locations (1):
- Leeds Teaching Hospitals NHS Trust, Leeds, United Kingdom